CLINICAL TRIAL: NCT02055742
Title: Clinical Study Protocol for the Illumigene® Chlamydia and Illumigene® Gonorrhea DNA Amplification Assays
Brief Title: Detection of Chlamydia (CT) and Gonorrhea (NG)
Status: Completed | Type: Observational
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MBI-01-CTNG; Meridian Bioscience, Inc. (Other: Meridian Bioscience, Inc.)
Record Dates: First submitted 2014-01-31; First posted 2014-02-05 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2014-09

CONDITIONS: Chlamydia; Gonorrhea
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Leftover urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Specimen Collection
  Interventions: Device: illumigene CT and NG assays, illumipro-10

INTERVENTIONS:
Device: illumigene CT and NG assays, illumipro-10

SUMMARY:
To evaluate the illumigene Chlamydia and illumigene Gonorrhea assays, using the illumipro-10, with male urine, female urine, physician-collected (medical professional) endocervical swabs and self-collected vaginal swabs taken from symptomatic and asymptomatic patient populations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Any ethnicity or race
3. Subject >14 and <89 years of age
4. Subject who voluntarily gives written informed consent; not applicable for leftover specimens
5. Symptomatic or asymptomatic subject who is able and willing to provide the required urine and swab samples for testing for CT and NG
6. Leftover urine specimens

Exclusion Criteria:

1. Subjects < 14 or >90 years of age
2. Subjects who are unwilling to sign the written informed consent; not applicable for leftover specimens
3. Subject who is unwilling or unable to provide the required urine and swab samples for testing; not applicable for leftover specimens
4. Individuals who have been on antibiotic medications within 10 days.
5. Multiple sets of specimens from the same subject at different office visits
6. Samples collected or processed in manner other than specified in the study protocol and Investigational Use Only package insert.
7. Frozen archived specimens

Ages: 14 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Symptomatic and asymptomatic subjects at least 14 years of age
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2014-03-01; Primary Completion 2014-09-09 (Actual); Study Completion 2014-09-09 (Actual)

PRIMARY OUTCOMES:
Qualitative detection of Chlamydia trachomatis and/or Neisseria gonorrhoeae (GC) to aid in the diagnosis of chlamydial and/or gonococcal urogenital disease | Up to 60 days
  Testing of each set of subject samples is completed within 60 days of sample collection

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Planned Parenthood of the Rocky Mountains, Aurora, Colorado
  - New England Center for Clinical Research, Fall River, Massachusetts
  - Planned Parenthood Southeastern PA, Philadelphia, Pennsylvania